CLINICAL TRIAL: NCT03385096
Title: Melphalan vs Busulfan+ Cyclophosphamide+ Etoposide Conditioning Regimen for Multiple Myeloma Undergoing Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Mel vs BUCY+VP-16 Conditioning Regimen for MM Undergoing Auto-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); Zhujiang Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mel vs BUCY+VP-16-MM-2017
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2019-02

CONDITIONS: Autologous Hematopoietic Stem Cell Transplantation; Conditioning; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Busulfan; Cyclophosphamide; Etoposide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUCY+VP-16 (Experimental): For MM patients undergoing auto-HSCT，BUCY+VP-16 conditioning regimen was BU 3.2 mg/kg/day on days -8 and -6；CY 60 mg/kg/day on days -5 and -4; VP-16 10mg/kg/day on days -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY); Drug: Etoposide (VP-16)
- Melphalan (Active Comparator): For MM patients undergoing auto-HSCT，Melphalan conditioning regimen was Melphalan 200mg/m2 on day -2.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -8 to -6.
  -7 to -4.
  Arms: BUCY+VP-16
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -5 to -4. on days -3 to -2.
  Arms: BUCY+VP-16
Drug: Etoposide (VP-16) — Etoposide was administered at 10 mg/kg/day on days -3 to -2.
  -3 to -2.
  Arms: BUCY+VP-16
Drug: Melphalan — Melphalan was administered at 200mg/m2 on day -2.
  Arms: Melphalan

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Melphalan and BUCY+VP-16 myeloablative conditioning regimens in multiple myeloma undergoing autologous hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma patients
* Achieving at least VGPR after chemotherapy, then mobilizing and collecting of peripheral blood stem cells

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
OS | 3 year
  overall survival (OS)

SECONDARY OUTCOMES:
relapse rate relapse rate | 3 year
  relapse rate
DFS | 3 year
  disease-free survival (DFS)
TRM | 3 year
  transplant-related mortality (TRM)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China